CLINICAL TRIAL: NCT07165132
Title: Phase 1 First-in-Human (FIH), Dose Escalation and Dose Expansion Study of RYZ401, a Novel Radiopharmaceutical Therapy Labeled With Actinium-225 (225Ac), in Subjects With Neuroendocrine Tumors (NETs) and Other Selected Solid Tumors Expressing Somatostatin Receptors (SSTRs).
Brief Title: Study of RYZ401 in Subjects With Solid Tumors Expressing SSTRs.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RYZ401-101
Record Dates: First submitted 2025-08-20; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: GEP-NET; Gastroenteropancreatic Neuroendocrine Tumor; Gastroenteropancreatic Neuroendocrine Tumor Disease; Neuroendocrine Tumors; Carcinoid; Carcinoid Tumor; Pancreatic NET; Solid Tumor; Somatostatin Receptor
Keywords: Neuroendocrine Tumors; SSTR+; GEP-NET; Targeted Radiotherapy; Gastroenteropancreatic Neuroendocrine Tumor; RayzeBio; Actinium; Ac 225; PRRT; Solid Tumor; Somatostatin Receptors; Radiopharmaceutical
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation, Dose Expansion (Experimental)
  Interventions: Drug: RYZ401

INTERVENTIONS:
Drug: RYZ401 — Ac-225

SUMMARY:
The primary objectives are to determine the recommended Phase 2 dose (RP2D) and optimal treatment regimen, characterize safety and tolerability, and evaluate preliminary efficacy of RYZ401 in subjects with NETs and other selected solid tumors expressing SSTRs.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years old at the time of signing the main study informed consent form (ICF).
* Histologically confirmed:

  * Grades 1-3 WD NETs (dose escalation and dose expansion)
  * Meningioma (dose expansion only)
* SSTR-positive disease, as assessed by SSTR-PET imaging
* Adequate renal, hematologic and hepatic function

Exclusion criteria:

* Prior RPT, including Lu-177.
* Prior solid organ or bone marrow transplantation.
* Use of chronic systemic steroid therapy.
* Significant cardiovascular disease
* Resistant hypertension
* Uncontrolled diabetes
* Prior history of liver cirrhosis
* HIV, hepatitis B infection or known active hepatitis C virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | Incidence of DLTs during the first 4 weeks of RYZ401 treatment
  Incidence of DLTs during RYZ 401 Treatment
Dose Expansion | Cycle1 Day 1 to LPFV + 6 weeks
  Incidence, severity, and duration of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Denis Ferreira, MD, Study Director — RayzeBio, Inc.